CLINICAL TRIAL: NCT02740244
Title: Effects of Intermittent Theta Burst Stimulation Applied Over the Left Dorsolateral Prefrontal Cortex in Patients With Treatment-resistant Bipolar Depression
Brief Title: Effect of Intermittent ThetaBurst Stimulation in Treatment-resistant Bipolar Depression
Acronym: iTBS-BIP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulties of recruitment
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 1018 rTMS DEP BIP
Record Dates: First submitted 2016-04-06; First posted 2016-04-15 (Estimated); Last update posted 2018-08-02 (Actual); Status verified 2018-07

CONDITIONS: Bipolar Depression
MeSH Terms: conditions — Bipolar Disorder | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- active iTBS (Active Comparator): Participants will receive 10 to 30 sessions of active intermittent theta burst stimulation (iTBS) consisting in delivering 2 s train of bursts containing three pulses at 50 Hz repeated each 200 ms every 10 s (iTBS). Each iTBS session contained 990 pulses and lasted 6 min. Stimulation intensity will be set at 80% of the patient's resting motor threshold. iTBS will be applied twice per day, with at least three hours between each session. Ten to 30 sessions will be delivered until patient achieved remission (i.e., 13-item Beck Depression Inventory (BDI13) score < 10). iTBS will be applied over the left dorsolateral prefrontal cortex (DLPFC) according to the individual's 3D-T1 MRI.
  Interventions: Device: active iTBS
- sham iTBS (Sham Comparator): The same protocol (location, intensity, parameters of stimulation) will be applied using a commercial sham coil.
  Interventions: Device: sham iTBS

INTERVENTIONS:
Device: active iTBS — Transcranial magnetic stimulation. MagProX100 (MagVenture, Denmark) with a figure-eight coil (MCF-B65)
  Other Names: intermittent Theta Burst stimulation; rTMS stimulator, rTMS
  Arms: active iTBS
Device: sham iTBS — Transcranial magnetic stimulation. MagProX100 (MagVenture, Denmark) with a sham figure-eight coil (MCF-P-B65)
  Other Names: sham intermittent Theta Burst stimulation; sham rTMS
  Arms: sham iTBS

SUMMARY:
The aim is to evaluate the evaluate the clinical interest and the safety of repetitive transcranial magnetic stimulation (rTMS) delivered as intermittent Theta burst stimulation(iTBS) on severity of depression in patients with treatment-resistant bipolar disorder.

DETAILED DESCRIPTION:
Methods: A double-blind randomized sham-controlled pilot study will be conducted in 40 patients with bipolar treatment-resistant depression receiving either active (n=20) or sham (n=20) iTBS over the left dorsolateral prefrontal cortex.

Depression severity will be assessed by an investigator blinded to iTBS condition before and after 10 to 30 iTBS sessions depending on remission onset. Remission will be defined as Beck Depression Inventory, BDI score<10.

Objective/Hypothesis: The investigators hypothesized the superiority of active iTBS over sham ITBS

ELIGIBILITY:
Inclusion Criteria:

* Bipolar disorder according to Diagnostic and Statistical Manual of Mental Disorders, DSM-IV criteria
* Montgomery and Asberg depression scale > 20

Exclusion Criteria:

* other psychiatric features, rapid cycles
* Benzodiazepines intake
* pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-01; Primary Completion 2011-02 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Beck Depression Inventory | 2 time point measure, before and after the end of stimulation sessions (changes from baseline BDI scores at 6 weeks)
  Self-reported clinical scale with 13 items

CONTACTS AND LOCATIONS:
Overall Officials: David Szekely, MD, Principal Investigator — University Hospital, Grenoble

IPD SHARING:
Plan to Share IPD: No